CLINICAL TRIAL: NCT00109668
Title: Evaluation of Two Doses of QVAR Versus Placebo by Breath Operated and Metered Dose Inhalers in Moderate Asthmatic Adolescents and Adults on a Stable Regimen of Inhaled Corticosteroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IXR-301-4-197
Record Dates: First submitted 2005-05-02; First posted 2005-05-03 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

INTERVENTIONS:
Drug: beclomethasone dipropionate (QVAR)

SUMMARY:
QVAR in a standard press and breath inhaler (QVAR-MDI) has been approved by the Food and Drug Administration (FDA) for use in the United States. The purpose of this study is to determine the level of asthma control when comparing the safety and effectiveness of QVAR in two different devices, a metered dose inhaler (MDI) and a breath operated inhaler (BOI).

DETAILED DESCRIPTION:
This investigation is a multicenter, randomized, placebo and active controlled, double-blind, double-dummy, parallel-group study to evaluate the safety and efficacy of two doses of QVAR-BOI in adolescents and adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female at least 12 years of age at the screening visit. NOTE: Females of childbearing potential may be included if they are practicing an acceptable method of contraception for at least 2 months and have a negative urine pregnancy test at the screening visit.
* Asthma (FEV1 60-85% predicted)
* Ability to perform acceptable and reproducible spirometry
* Ability to perform PEF determinations
* Reversible bronchoconstriction as verified by a greater than or equal to 12% increase in FEV1 following inhalation of albuterol. Historical reversibility will be allowed
* Patients must be on a stable regimen of daily-inhaled corticosteroids at low to medium doses for at least 30 days prior to screening.
* Otherwise healthy individuals with clinically-acceptable medical history, physical examination, vital signs, 12 lead ECG, and clinical laboratory parameters within the acceptable ranges for asthma patients.
* Non-smoker for at least one year prior to the screening visit and maximum smoking history of ten-pack years
* The patient must be willing to give written informed consent and be able to adhere to the dose and visit schedules. If applicable, parent or guardian must also provide consent.

Exclusion Criteria:

* Allergy or sensitivity to BDP (beclomethasone dipropionate) or to other components of the formulations used in the CTM
* Patients demonstrating an increase or decrease in FEV1 >20% between the screening and baseline visit.
* Patients requiring the use of >12 puffs per day of albuterol for any 3 consecutive days between the screening and baseline visits.
* Patients who are unable to use an MDI without a spacer device. (Use of spacers is prohibited during the course of the study.)
* Patients who have been treated with methotrexate, cyclosporin, gold or other cytotoxic agents for the control of asthma or for a concurrent condition within the last 3 months.
* Patients who are receiving escalating doses of immunotherapy, oral immunotherapy or short course (rush) immunotherapy for rhinitis.
* Patients with evidence of oropharyngeal candidiasis.
* Exposure to investigational drugs within 30 days prior to the screening visit
* Require continuous treatment with beta blockers (administered by any route), MAO inhibitors, leukotriene modifiers, tricyclic antidepressants, anticholinergics, inhaled nedocromil or cromolyn, or nebulized therapy (excluding sponsor provided albuterol MDI) following the screening visit.
* Patients who have received any of the following treatments or met any of the following conditions within six weeks prior to the screening visit: *oral or injectable corticosteroids; *an upper respiratory tract infection and/or sinusitis associated with exacerbation of asthmatic symptoms; *emergency room treatment or hospitalization for asthmatic symptoms
* Inability to tolerate or unwillingness to comply with required washout periods for all applicable medications
* Treatment at any time for life-threatening asthmatic episodes
* History or presence of any non-asthmatic acute or chronic lung disease
* History of glaucoma, ocular hypertension or cataracts
* Presence of systemic fungal, bacterial, viral or parasitic infections and/or ocular herpes simplex
* Known or suspected substance abuse (e.g., alcohol, marijuana, etc.)
* Patients who are known to be HIV positive
* Unlikely to be compliant, take study medication as directed, complete the diary cards, or attend scheduled clinic visits as required.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 415
Dates: Start 2004-07-31 (Actual); Primary Completion 2006-09-30 (Actual); Study Completion 2006-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (31):
  - Alabama Allergy and Asthma, Birmingham, Alabama
  - Allergy and Asthma Specialists, Huntington Beach, California
  - West Coast Clinical Trials, Long Beach, California
  - Allergy Research Foundation, Los Angeles, California
  - UCLA David Geffen School of Medcine, Los Angeles, California
  - Clinical Trials of Orange County, Inc., Orange, California
  - Allergy Associates Medical Group, San Diego, California
  - Allergy and Asthma Medical Group, Walnut Creek, California
  - Boulder Medical Center, Boulder, Colorado
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Center, Denver, Colorado
  - Asthma and Allergy Research Center, Sarasota, Florida
  - Allergy and Asthma DTC, Tallahassee, Florida
  - Aero Allergy Research Labs of Savannah, Inc, Savannah, Georgia
  - Pulmonary Consultants of North Idaho, Coeur d'Alene, Idaho
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Family Allergy and Asthma Research Center, Louisville, Kentucky
  - Bendel Medical Research, Lafayette, Louisiana
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - The Clinical Research Center, St Louis, Missouri
  - Dr. Alan Kaufman, The Bronx, New York
  - Regional Allergy and Asthma Consultants, Asheville, North Carolina
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy, Asthma & Dermatology Research Center, Lake Oswego, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - National Allergy and Asthma and Urticaria Centers of Charleston, PA, Charleston, South Carolina
  - Allergy and Asthma Associates, Houston, Texas
  - Dr. Emory Robinette, Abingdon, Virginia
  - Belligham Asthma and Allergy, Bellingham, Washington
  - Pulmonary Consultants, Tacoma, Washington
  - Morgantown Pulmonary Associates, Morgantown, West Virginia
- Ponce School of Medicine, Ponce, Puerto Rico